CLINICAL TRIAL: NCT02449811
Title: Single-center, Randomized, Open-label, Parallel-group Study to Characterize Renin-angiotensin-system (RAS) Peptide Profiles Before and After Treatment Initiation With Different Antihypertensive Drug-classes in Patients With Treatment-naive Arterial Hypertension
Brief Title: RAS Peptide Profiles in Patients With Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2015-081
Record Dates: First submitted 2015-04-10; First posted 2015-05-20 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Perindopril; olmesartan; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Perindopril: Treatment period 1: Perindopril 5mg, oral, once daily, for 4 weeks Treatment period 2: Perindopril 10mg, oral, once daily, for 4 weeks
  Interventions: Drug: Perindopril
- Olmesartan: Treatment period 1: Olmesartan 20mg, oral, once daily, for 4 weeks Treatment period 2: Olmesartan 40mg, oral, once daily, for 4 weeks
  Interventions: Drug: Olmesartan
- Amlodipine: Treatment period 1: Amlodipine 5mg, oral, once daily, for 4 weeks Treatment period 2: Amlodipine 10mg, oral, once daily, for 4 weeks
  Interventions: Drug: Amlodipine
- Hydrochlorothiazide: Treatment period 1: Hydrochlorothiazide 25mg, oral, once daily, for 4 weeks Treatment period 2: Hydrochlorothiazide 50mg, oral, once daily, for 4 weeks
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Perindopril
  Groups: Perindopril
Drug: Olmesartan
  Groups: Olmesartan
Drug: Amlodipine
  Groups: Amlodipine
Drug: Hydrochlorothiazide
  Groups: Hydrochlorothiazide

SUMMARY:
Randomized, open-label, parallel-group study conducted at a single center in Switzerland.

Patients diagnosed with primary arterial hypertension requiring antihypertensive drug Treatment as well as patients after a 4 week wash out period (Amendment 07/2016) will be recruited at the University Hospital Basel, Switzerland. Subjects will be randomized to either the angiotensin-converting enzyme inhibitor-, angiotensin receptor blocker-, calcium channel blocker- or hydrochlorothiazide-treatment arm. Drug treatment follows current guidelines issued by the European Society of Hypertension. Treatment-naive patients will be started on an intermediate dose monotherapy (treatment period 1). In all patients who do not reach blood pressure targets after 4 weeks, the dose of the monotherapy drug will be doubled (high dose, treatment period 2). Sampling for the analysis of RAS peptide profiles, measurement of drug concentrations in plasma and non-invasive hemodynamic measurements will be done. A control group with 20 age and gender matched, healthy and normotensive subjects will be recruited to establish the characteristics of the RAS peptide profiles in a comparable but normotensive population.

DETAILED DESCRIPTION:
This will be a single-center, randomized, open-label, parallel-group study in patients with treatment-naive arterial hypertension to characterize RAS peptide profiles before and after treatment initiation with different antihypertensive drug-classes. Patients diagnosed with primary arterial hypertension requiring antihypertensive drug treatment as well as patients after a 4 week wash out period (Amendment from 07/2016) will be recruited from the Medical Outpatient Clinic at the University Hospital Basel, Switzerland. Diagnostic work-up and follow-up assessments after treatment initiation such as 24 hour blood pressure measurement will be performed according to clinical practice guidelines and will only be documented but not altered by this study. Study mandated procedures will be randomization to one of the four standard first-line treatment arms, blood sampling for RAS peptide profile and drug concentration determination, and non-invasive hemodynamic measurements. After having provided written informed consent, patients will be randomized to either the angiotensin-converting enzyme inhibitor-, angiotensin receptor blocker-, calcium channel blocker- or hydrochlorothiazide-treatment arm. Drug treatment follows current guidelines issued by the European Society of Hypertension . According to clinical practice, treatment-naive patients with grade I and grade II hypertension will directly be started on an intermediate dose monotherapy (treatment period 1).

Treatment period 1:

4 weeks of intermediate dose monotherapy with the angiotensin-converting enzyme Inhibitor perindopril OR the angiotensin receptor blocker olmesartan OR the calcium channel blocker amlodipine OR the hydrochlorothiazide

In all patients who do not reach blood pressure targets according to the 2013 ESH guidelines for the management of arterial hypertension after 4 weeks, the dose of the monotherapy drug will be doubled (high dose, treatment period 2), following current guidelines

Treatment period 2:

4 weeks of high dose monotherapy with the angiotensin-converting enzyme inhibitor perindopril OR the angiotensin receptor blocker olmesartan OR the calcium channel blocker amlodipine OR the hydrochlorothiazide

80 patients (20 patients per treatment arm) will be included and sampling for the analysis of RAS peptide profiles will be done before treatment initiation (baseline). Sampling for the analysis of RAS peptide profiles and measurement of drug concentrations in plasma will be done after 4 weeks of each treatment period at 0h (before last drug intake) and 4 hours after last drug intake of treatment period. Dropouts will be replaced. Non-invasive hemodynamic measurements will be done at the same time points as for the determination of RAS peptide profiles and drug concentrations.

A control group with 20 age- and gender-matched, healthy and normotensive subjects will be recruited to establish the characteristics of RAS peptide profiles in a comparable but normotensive population. After having provided written informed consent, normal blood pressure will be documented by a 24h blood pressure measurement. In this normotensive control group, blood sampling for the determination of RAS peptide profiles as well as hemodynamic measurements will only be done on a single day, at the same time of day as for the hypertensive patients. (Amendment 04/2015)

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients with previously untreated non-secondary arterial hypertension, defined as: office-systolic blood pressure ≥ 140 mmHg and ≤ 180 mmHg and office-diastolic blood pressure ≥ 90 mmHg and ≤110 mmHg (ESH grade I and II hypertension).
* Male or female outpatients with previously treated non-secondary arterial Hypertension after a wash out period of 4 weeks (Amendment 07/2016)
* Evaluation of 24h blood pressure measurement fulfills criteria of hypertension: mean systolic blood pressure / diastolic blood pressure ≥ 130/80 on average, ≥ 135/85 during the day, or ≥ 120/70 during the night.
* Age ≥ 18 years
* Body mass index between 18 and 35 kg/m²
* Body weight at least 50 kg
* Ability to understand study procedures and to provide written informed consent
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening.
* 12-lead ECG without clinically relevant abnormalities (Exception: signs of left ventricular hypertrophy with Sokolow index >3.5mV).
* Female study participants less than one year post-menopausal must, be non-pregnant and non-lactating, and willing to use an adequate and highly effective method of contraception throughout the study and for 1 week after the last dose. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as, implants, injectables, combined oral contraceptives, some intrauterine devices (IUD) (hormonal) in combination with a condom or sterilisation, sexual abstinence or vasectomised partner.

Exclusion Criteria:

* Pregnant or lactating women
* Clinical chemistry results indicating secondary arterial hypertension.
* History of or clinically evident cardiovascular disease (other than arterial hypertension), namely myocardial infarction and valvular heart disease or heart failure.
* Ventricular or dual pacemaker wearers
* Uni- or bilateral renal artery stenosis
* Renal dysfunction, defined as estimated creatinine-clearance < 60 ml/min
* Recipient of kidney transplant
* Moderate or severe hepatic impairment
* Clinically relevant lung disease (e.g. uncontrolled bronchial asthma, chronic obstructive pulmonary disease (COPD))
* History of alcohol abuse
* Loss of ≥ 250 ml of blood within 3 months prior to screening.
* Known hypersensitivity to any of the four antihypertensive drugs or any excipients of the drug formulations
* History or clinical evidence of any disease and / or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity.
* Participation in another clinical trial within past 30 days
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
RAS peptide profiles | 0h and 4h
  Concentration measurement of the different RAS peptides

SECONDARY OUTCOMES:
Composite measure of Non-invasive hemodynamic parameters | 0h and 4h
  Composite measure of Non-invasive hemodynamic parameters to include: Cardiac index, Stroke index, Mean arterial pressure, Ejection phase contractility index, Inotropic state index, Left stroke work index, Stroke systemic vascular resistance index, Thoracic fluid conductivity
Plasma renin activity and aldosterone concentration | 0h and 4h
Antihypertensive drug concentrations | 0h and 4h

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, Prof. Dr. med., Principal Investigator — University of Bern
Locations (1):
- University Hospital, Basel, Switzerland